CLINICAL TRIAL: NCT00921648
Title: Xijing HOSPITAL, Fourth Military Medical University, China
Brief Title: Clinical Findings in General Paresis
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Department of neurology, xijing hospital
Other Study IDs: 20080301
Record Dates: First submitted 2008-10-21; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: General Paresis
Keywords: EEG; general paresis; MRI; neurosyphilis
MeSH Terms: conditions — Neurosyphilis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Mr Q, 40 years old: Dementia, sensory aphasia, irritability, hallucination MRI showed cortical lesion, mesial temporal lobe atrophy.
- Mr Guo,35 years old: Dementia, sensory aphasia, tremor, gait disturbance MRI showed cortical lesion, enlarged ventricle, white matter lesion, cerebral atrophy
- Mr Zhang,40 years old: Dementia, apraxia of speech, gatism , irritability, insomnia, gait disturbance MRI showed white matter lesion, cerebral atrophy.
- Mr Liu,40 years old: Dementia, apraxia of speech, irritability, insomnia MRI showed normal.
- Mr Zhang,54 years old: Dementia, apraxia of speech MRI showed white matter lesion, cerebral atrophy.

SUMMARY:
This is a study of the clinical and neuroimaging of general paresis. The investigators studied six patients with general paresis.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Mental disorders
* positive TPHA in CSF and sera
* HIV-negative serology by ELISA

Exclusion Criteria:

* Negative TPHA in CSF and sera
* No image data

ELIGIBILITY:
Inclusion Criteria:

* EEG MR

Exclusion Criteria:

* Serological test

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 6 cases
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: yuangui huang, MD, Study Director — department of neurology ,xijing hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China